CLINICAL TRIAL: NCT00433316
Title: Pain Relief by Continuous Intra-Peritoneal Nebulization of Ropivacaine During Gynecological Laparoscopic Surgery
Brief Title: Pain Relief by Intra-Peritoneal Ropivacaine During Gynecological Laparoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Yuval Kaufman, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMC064113CTIL; HT 3758
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2007-02

CONDITIONS: Laparoscopic Surgical Procedures
Keywords: ropivacaine; laparoscopy; intraperitoneal; nebulization; pain; local analgesic; gynecology
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study (Experimental): Receiving 10ml of 1% ropivacaine
  Interventions: Drug: ropivacaine
- Control (Placebo Comparator): Receiving 10ml of saline
  Interventions: Device: Aeroneb Pro Nezulizer, Aerogen, Ireland

INTERVENTIONS:
Drug: ropivacaine — 1% ropivacaine
  Other Names: Narop
  Arms: study
Device: Aeroneb Pro Nezulizer, Aerogen, Ireland — Aeroneb Pro Nezulizer, Aerogen, Ireland
  Arms: Control

SUMMARY:
In our prospective, randomized, placebo controlled and double-blinded study we will study the efficacy of intraperitoneal ropivacaine nebulization on pain relief during gynecological laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective gynecologic laparoscopic surgery including unilateral or bilateral salpingo-oopherectomy or ovarian cystectomy.
* The patient is not participating in other medical study at present or in the last 30 days.
* The patient signed on an informed consent.
* Age 18 years and above.
* ASA (American Society of Anesthesiologists) physical status grade 1- 2.

Exclusion Criteria:

* Allergy to Ropivacaine, other local anesthetics or other medications listed in the protocol.
* The patient is participating in other medical experiment at present or in the last 30 days.
* Acute Pelvic Inflammatory Disease.
* Coumadin or Aspirin treatment.
* ASA physical status grade 3-4.
* Age < 18 years.
* Significant arrythmias
* Analgesic treatment for chronic pain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
VAS score | early post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Kaufman, MD, Principal Investigator — Carmel Medical Center, Haifa, Israel; Reuven Pizov, Prof., Study Director — Carmel Medical Center, Haifa, Israel
Locations (1):
- the Carmel Medical Center Ambulatory Gynecoendoscopic Unit, Haifa, Israel